CLINICAL TRIAL: NCT02267980
Title: Turgut Ozal Medical Center Department of Anesthesiology and Reanimation
Brief Title: Effect of the Addition of Ketamine to Sevoflurane Anesthesia in Electroconvulsive Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Feray Erdil, Associated Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inonu 2
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Depressive Disorder
Keywords: Electroconvulsive therapy; sevoflurane; ketamine
MeSH Terms: conditions — Depressive Disorder | interventions — Sevoflurane; Ketamine; Injections; Sodium Chloride; Isotonic Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group SK (Active Comparator): Sevoflurane was initiated, in both groups, at 8% for anesthesia induction until loss of consciousness was achieved, at which point it was discontinued. Following loss of consciousness ketamine was administered to Group SK (n=29) in the form of a 0.5mg/kg iv bolus. Patients in Group SS (n=30) received saline in the same manner.
  Interventions: Drug: Sevoflurane; Drug: Ketamine
- Group SS (Placebo Comparator): Sevoflurane was initiated, in both groups, at 8% for anesthesia induction until loss of consciousness was achieved, at which point it was discontinued. Patients in Group SS (n=30) received saline in the same manner.
  Interventions: Drug: Sevoflurane; Drug: Saline

INTERVENTIONS:
Drug: Sevoflurane — Inhalation anesthetic agent
  Other Names: Sevoflurane (sevorane)
Drug: Ketamine — Intravenous anesthetic agent
  Other Names: Ketamine (Ketalar) 50mg/mL injection
  Arms: Group SK
Drug: Saline — Isotonic solution for placebo group
  Other Names: Isotonic solution
  Arms: Group SS

SUMMARY:
The investigators evaluate the effects of a subanesthetic dose of ketamine, administered as an adjunct to sevoflurane, on duration of seizure activity, hemodynamic profile and recovery times during electroconvulsive therapy (ECT) in patients with major depression.

DETAILED DESCRIPTION:
Patients will randomly allocate, to either a sevoflurane-ketamine (Group SK), sevoflurane-saline (Group SS) receiving group. Mean arterial pressure (MAP) and heart rate (HR) will record prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 min after the seizure has ended (T3, T4, T5, and T6, respectively). Motor and EEG seizure durations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive patients

Exclusion Criteria:

* Pregnancy
* Have a history of myocardial infarction in the previous six months
* Atrial fibrillation or flutter
* Heart block
* Unregulated hypertension
* Cerebrovascular diseases
* A known drug allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
seizure duration | During electroconvulsive therapy (30 minutes)
  the time from application of the ECT stimulus to the cessation of tonic-clonic motor activity in the isolated arm.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | During Electroconvulsive therapy (30 minutes)
  Mean arterial pressure (MAP) will be recorded prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 min after the seizure has ended (T3, T4, T5, and T6, respectively).
Heart rate (HR) | During Electroconvulsive therapy (30 minutes)
  Heart rate (HR) will be recorded prior to anesthetic induction (T1); following anesthetic induction (T2); and 0, 1, 3, and 10 min after the seizure has ended (T3, T4, T5, and T6, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Feray Erdil, MD, Principal Investigator — MD
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Yalcin S, Aydogan H, Selek S, Kucuk A, Yuce HH, Karababa F, Bilgic T. Ketofol in electroconvulsive therapy anesthesia: two stones for one bird. J Anesth. 2012 Aug;26(4):562-7. doi: 10.1007/s00540-012-1378-6. Epub 2012 May 24. PMID 22623080